CLINICAL TRIAL: NCT00594620
Title: A Prospective Trial of Soy Derivatives for Control of Hot Flashes in Men on Androgen Deprivation Therapy
Brief Title: Soy Derivatives for Control of Hot Flashes in Men on Androgen Deprivation Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to poor accrual and without sufficient patients or data to report on any outcomes.
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 9639
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Results first posted 2022-02-08 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Subjects receive supplement
  Interventions: Dietary Supplement: Flav-ein capsules
- 2 (Placebo Comparator): Subjects will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Flav-ein capsules — Soy/isoflavone supplementation
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
To determine the efficacy of soy/isoflavone supplementation on hot flashes in men who are being treated with luteinizing hormone-releasing hormone (LHRH) agonist therapy for control of advanced prostate cancer

DETAILED DESCRIPTION:
Literature has shown that low dose estrogens can control hot flashes in men on androgen deprivation but with a high risk of thromboembolic events. Soy derivatives that contain isoflavones, a type of phytoestrogen, have been evaluated in peri-menopausal women as a possible safer alternative to synthetic estrogens but there has not been a similar study performed on their effect in men on androgen deprivation therapy for prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of prostate with treatment of prostate cancer (radical prostatectomy, radiation therapy, etc.)
* had biochemical/clinical relapse and started on antiandrogens
* have documented history of hot flashes

Exclusion Criteria:

* History of MI, DVT, CVA
* peanut allergy
* untreated hypothyroidism
* must be off other medical treatment for hot flashes for 2 weeks before enrollment in this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2004-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M. Holzbeierlein, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was terminated early due to low accrual. Study was blinded and no data was collected
Groups:
- Arm 1/ Soy Supplementation: Subjects receive supplement
  Flav-ein capsules: Soy/isoflavone supplementation
- Arm 2/ Placebo: Subjects will receive placebo
  Placebo: Placebo
Period: Overall Study
Arm/Group | Arm 1/ Soy Supplementation | Arm 2/ Placebo
Started | 0 (Study was terminated early due to low accrual. Study was blinded and no data was collected) | 0 (Study was terminated early due to low accrual. Study was blinded and no data was collected)
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This trial was stopped early due to low enrollment. There was not a sufficient number of participants to accurately analyze the data. Randomization was not completed prior to termination. Data for population analysis not collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1/ Soy Supplementation | Arm 2/ Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Ethnicity (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Using Isoflavones as Safer Alternative to Synthetic Estrogens
Time Frame: 16 Weeks
Population: The trial was stopped early due to failure to accrue Not enough subjects were enrolled with enough follow up to have data
Groups:
- Flav-ein Capsules: Subjects receive supplement
  Flav-ein capsules: Soy/isoflavone supplementation
- Placebo: Subjects will receive placebo
  Placebo: Placebo
Arm/Group | Flav-ein Capsules | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Flav-ein Capsules | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

LIMITATIONS AND CAVEATS:
Early termination due to low accrual. Insufficient number of participants for accurate analysis. No data collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes